CLINICAL TRIAL: NCT00510913
Title: Prograf® (Tacrolimus) as Secondary Intervention vs. Continuation of Cyclosporine in Patients at Risk for Chronic Renal Allograft Failure
Brief Title: A Study to Compare the Conversion to Prograf® (Tacrolimus) to the Continuation of Cyclosporine in Patients at Risk for Chronic Renal Allograft Failure
Acronym: CRAF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20-98-002
Record Dates: First submitted 2007-07-31; First posted 2007-08-02 (Estimated); Last update posted 2007-08-02 (Estimated); Status verified 2007-07

CONDITIONS: Graft Rejection; Kidney Transplantation
Keywords: Treatment efficacy; Transplantation rejection; Kidney transplantation; Cyclosporine; tacrolimus
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: tacrolimus
  Other Names: Prograf®, FK506

SUMMARY:
A study to compare the conversion to Prograf® (tacrolimus) to the continuation of cyclosporine in patients at risk for chronic renal allograft failure

DETAILED DESCRIPTION:
A two arm study (1 Active, 1 Active control) to compare the incidence, progression and severity of chronic renal allograft failure in at-risk patients who are converted from cyclosporine-based to tacrolimus-based immunosuppression to patients who remain on cyclosporine-based therapy

ELIGIBILITY:
Inclusion Criteria:

* Patient has been on cyclosporine-based immunosuppression regimen since the transplant
* Patient has at least one pre-defined risk factor for chronic allograft failure

Exclusion Criteria:

* Patient is dialysis dependent
* Patient is recipient of a solid organ transplant other than the kidney

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 1999-02; Study Completion 2000-09 (Actual)

PRIMARY OUTCOMES:
Graft Survival | 5 years

SECONDARY OUTCOMES:
Patient survival, Graft Loss | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: John Holman, MD, Study Director — Astellas Pharma Inc
Locations (18):
- United States (18):
  - Los Angeles, California
  - San Diego, California
  - San Francisco, California
  - Denver, Colorado
  - New Haven, Connecticut
  - Augusta, Georgia
  - Chicago, Illinois
  - Lexington, Kentucky
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Minneapolis, Minnesota
  - Albany, New York
  - New York, New York
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Nashville, Tennessee
  - Salt Lake City, Utah
  - Madison, Wisconsin